CLINICAL TRIAL: NCT01650727
Title: A Phase 1b Trial of Dinaciclib in Combination With Rituximab in Subjects With Relapsed and Refractory Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma
Brief Title: A Study of Dinaciclib in Combination With Rituximab in Participants With Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma (P07974)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P07974; 2012-001437-14 (EudraCT Number); MK-7965-011 (Other: Merck Study Number)
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — dinaciclib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dinaciclib + Rituximab (Experimental): Rituximab will be administered in Cycles 1 and 3-13.
  Dinaciclib will be administered in Cycles 2-13.
  Interventions: Drug: Dinaciclib; Biological: Rituximab

INTERVENTIONS:
Drug: Dinaciclib — Dinaciclib is given as a single intravenous (IV) dose on Days 1, 8, and 15 in Cycle 2 through Cycle 13 (28 day cycles) at a starting dose of 7 mg/m^2 up to a maximum dose of 14 mg/m^2.
  Other Names: SCH 727965; MK-7965
Biological: Rituximab — Rituximab 375 mg/m^2 will be administered IV on Day 1, 8, 15 and 22 in Cycle 1 (28 day cycle) and on Day 1 in Cycles 3-13 (28 day cycles).
  Other Names: Rituxan®

SUMMARY:
The purpose of this study is to determine the maximum-tolerated dose (MTD) of dinaciclib therapy in combination with rituximab in chronic lymphocytic leukemia (CLL) and small lymphocytic lymphoma (SLL).

ELIGIBILITY:
Inclusion Criteria:

* Must have received at least one prior therapy that includes either

fludarabine or equivalent nucleoside analogue or an alternative regimen

* Diagnosis of chronic lymphocytic leukemia (CLL) or small lymphocytic

lymphoma (SLL)

* Eastern Cooperative Oncology Group (ECOG) Performance status ≤ 2
* Women of child-bearing potential who are sexually active, ,including both female subjects and the female sexual partners of male subjects, must agree to use a medically accepted method of contraception prior to enrollment, while receiving protocol-specified treatment, and for 12 months after stopping study treatment.
* Women of child-bearing potential who are not currently sexually active must

agree to use a medically accepted method of contraception should they become

sexually active while participating in the study.

* Life expectancy ≥12 weeks

Exclusion Criteria:

* Symptomatic brain metastases or primary central nervous system malignancy
* Treatment with any chemotherapy or biologic therapy within 4 weeks prior to enrollment
* Non-hematological toxicities from prior therapy
* Presence of any serious or uncontrolled infection defined as infection requiring hospital admission and/or parenteral antibiotics
* Known human immunodeficiency virus (HIV) infection or a known HIV-related

malignancy

* Clinically active hepatitis B or C defined as disease that requires

therapy

* Women who are breast-feeding, pregnant, or intend to become pregnant
* Prior allogeneic bone marrow transplant (auto hematopoietic stem cell

transplantation [HSCT] is allowed if fully recovered)

* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer or other cancer from which the subject is

considered by his or her physician to have a 2 year survival expectation

* Any investigational drugs within 4 weeks prior to the start of treatment
* Concurrently receiving treatment in any other clinical study
* Previously treated with a cyclin dependent kinase (CDK) inhibitor (e.g., dinaciclib or flavopiridol)
* Active autoimmune anemia or idiopathic thrombocytopenic purpura (ITP) unless

stable, defined as being responsive to corticosteroids or other standard therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing a Dose Limiting Toxicity (DLT) | Cycles 2 & 3 (Days 29-84)

REFERENCES:
- [Result] Fabre C, Gobbi M, Ezzili C, Zoubir M, Sablin MP, Small K, Im E, Shinwari N, Zhang D, Zhou H, Le Tourneau C. Clinical study of the novel cyclin-dependent kinase inhibitor dinaciclib in combination with rituximab in relapsed/refractory chronic lymphocytic leukemia patients. Cancer Chemother Pharmacol. 2014 Nov;74(5):1057-64. doi: 10.1007/s00280-014-2583-9. Epub 2014 Sep 13. PMID 25217392